CLINICAL TRIAL: NCT00770302
Title: An Open Label, Pharmacokinetic Study of Single and Multiple Doses of 5 mg Saxagliptin in Healthy Chinese Subjects Living in China
Brief Title: Assess Pharmacokinetics, Safety and Tolerability in Healthy Chinese Volunteers After Oral Doses of Saxagliptin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Peter Öhman, MD, PhD, Medical Science Director, AstraZeneca Pharmaceuticals
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D1680C00004
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Last update posted 2009-07-09 (Estimated); Status verified 2009-07

CONDITIONS: Type 2 Diabetes
Keywords: DPP-4 inhibitors; HBA1c; Incretins; Pharmacokinetics
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — saxagliptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Saxagliptin — Oral tablet, once daily for 1 (single-dose) and 5 (multiple-dose) days
  Other Names: ONGLYZA™

SUMMARY:
Saxagliptin is a new investigational medication being developed for treatment of type 2 diabetes. This Phase I study is designed to assess the pharmacokinetics of saxagliptin and its pharmacologically active metabolite, BMS-510849, following single and multiple oral doses of 5 mg saxagliptin in healthy Chinese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Men or women (not of childbearing potential) of Chinese ethnicity
* Weigh at least 50 kg and have a body mass index (BMI) between 19 and 24 kg/m2
* Must have normal physical examination, laboratory values, ECG, pulse and blood pressure unless the investigator considers an abnormality to not be clinically significant.

Exclusion Criteria:

* History of clinically significant hypoglycaemia (low blood sugar levels)
* Women who are pregnant or breastfeeding

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2008-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic variables for saxagliptin after single and multiple oral doses of 5 mg saxagliptin | Multiple timepoints during 9 days

SECONDARY OUTCOMES:
Pharmacokinetic variables for saxagliptin's active metabolite BMS-510849 after single and multiple oral doses of 5 mg saxagliptin | Multiple time points during 9 days
Safety variables (adverse events reported, vital sign measurements, electrocardiograms, physical examinations, and clinical laboratory tests after single and multiple oral doses of 5 mg saxagliptin | Multiple time points during 10 days (including measurements before dosing)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Öhman, MD, PhD, Study Director — AstraZeneca; Deborah Price, MSc, Study Chair — AstraZeneca
Locations (1):
- Research Site, Beijing, China

REFERENCES:
- [Derived] Li H, Yang L, Tou CK, Patel CG, Zhao J. Pharmacokinetic study of saxagliptin in healthy Chinese subjects. Clin Drug Investig. 2012 Jul 1;32(7):465-73. doi: 10.2165/11598760-000000000-00000. PMID 22668067